CLINICAL TRIAL: NCT02748382
Title: Fluids in Sepsis and Septic Shock: A Pilot Randomized Controlled Trial
Brief Title: Fluids in Sepsis and Septic Shock
Acronym: FISSH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1636
Record Dates: First submitted 2016-04-08; First posted 2016-04-22 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- higher chloride solutions (Active Comparator): higher chloride crystalloid (Normal saline) higher chloride albumin (5% Octalbin)
  Interventions: Other: higher chloride crystalloid; Other: higher chloride albumin
- lower chloride solutions (Active Comparator): lower chloride crystalloid (Ringer's lactate) lower chloride albumin (5% Plasbumin)
  Interventions: Other: lower chloride crystalloid; Other: lower chloride albumin

INTERVENTIONS:
Other: higher chloride crystalloid — Normal saline
  Arms: higher chloride solutions
Other: higher chloride albumin — 5% Octalbin
  Arms: higher chloride solutions
Other: lower chloride crystalloid — Ringers Lactate
  Arms: lower chloride solutions
Other: lower chloride albumin — 5% Plasbumin
  Arms: lower chloride solutions

SUMMARY:
Despite evidence of the physiologic benefits and possible lower mortality associated with low chloride solutions, normal saline remains the most wildly used fluid in the world. Given uncertainty about the impact of lower chloride versus higher chloride solutions on mortality, it is unlikely that clinical practice will change without new and direct RCT evidence. Editorials published in leading critical care journals have called for RCT's to address this important clinical question. The proposed feasibility RCT will investigate the feasibility of a large-scale trial directly comparing low chloride versus normal chloride for resuscitation in septic shock on patient-important outcomes such as mortality and AKI.

DETAILED DESCRIPTION:
Severe infection can lead to many complications within the human body including low blood pressure, which is called septic shock. The main treatments for septic shock are intravenous antibiotics and intravenous fluid.

There are many different intravenous fluids available for doctors to use. Each one of these fluids has potential advantages as well as potential disadvantages. Doctors will often look at many things when deciding which fluid to give including the results of bloodwork and the clinical characteristics of the patients themselves. There is limited direction from research studies taht using one fluid type is better than another. Some preliminary research in the field has suggested that one specific electrolyte, call chloride, may be harmful when given to patients in high concentrations. Animal research has shown that the administration of high chloride fluids may be harmful to the lungs, kidneys, gastrointestinal and muscle cells. Some intravenous fluids have higher concentrations of chloride than others.

The investigators plan to study the impact of giving patients with severe infection intravenous fluids with either a high chloride concentration (normal saline or high chloride albumin) or a low chloride concentration (Ringers Lactate or low chloride albumin). Although, the investigators plan for a larger trial looking at patient-important outcomes such as rate of death, kidney failure and length of stay in the ICU the investigators think it's important to start with a feasibility study. If the investigators are able to show a larger trial is feasible then the investigators will apply for further funding and use the lessons learned from this pilot to optimize the larger study. The larger study has the potential to guide the care of critically ill patients with infection worldwide.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 16 years of age
2. Within 6 hours from presentation to hospital or activation of MET/RACE team to ward
3. Requires fluid resuscitation for refractory hypotension OR organ hypoperfusion

   * refractory hypotension definition - sBP <90 OR MAP <65 after 1L bolus given over 1 hour or less
   * organ hypoperfusion - lactate >4
4. Suspected source of infection as etiology for hypotension
5. Treating physician anticipates patient will require admission to ICU

Exclusion Criteria:

1. Intracranial bleed or intracranial hypertension during this hospital admission
2. Acute burn injury (>10% body surface area)
3. Bleeding/hemorrhage as likely cause of hypotension
4. Plan in place to change goals of care to palliation
5. Previously enrolled in FISSH
6. Previously enrolled in confounding trial
7. Transfer from another hospital or facility
8. Admission directly from the operating room or PACU

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2017-08-19 (Actual); Study Completion 2017-08-19 (Actual)

PRIMARY OUTCOMES:
Consent Rate | 12 months
  Consent rate will be considered adequate if greater than 70% of substitute decision makers (SDMs) or patients when approached for consent choose to participate.
Patient Recruitment | 12 months
  Successful recruitment will be defined as achieving enrolment of 50 patients over the 12-month study period. This works out to approximately 1 patient/center/month. Once the pilot trial begins, the screening logs will be reviewed at all three study centers by the study steering committee on a monthly basis. We will record exclusions and reasons for physician refusals.
Protocol Adherence | 12 months
  Successful adherence will be defined as patients receiving at least 75% study fluid of all intravenous fluid that is administered in the ICU excluding blood products and medication infusions.

SECONDARY OUTCOMES:
Hospital length of stay | Duration of index hospital stay censored at 90 days.
Hospital mortality | hospital stay or up to 90 days
  Mortality during index hospitalization censored at 90 days.
Renal replacement therapy use | RRT use during index hospital stay censored at 90 days.
  Any use of renal replacement therapy including hemodialysis, peritoneal dialysis or continuous renal replacement. This will be reported as a dichotomous outcome.
ICU length of stay | Duration of index ICU stay censored at 90 days.
Hyperkalemia | Incidence during index ICU stay or up to 30 days
  Number of participants with any serum potassium value >5mmol/L.
Acidosis | Incidence during index ICU stay or up to 30 days
  Number of participants with any serum pH <7.20

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Juravinski Hospital-Hamilton Health Sciences, Hamilton, Ontario
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rochwerg B, Millen T, Austin P, Zeller M, D'Aragon F, Jaeschke R, Masse MH, Mehta S, Lamontagne F, Meade M, Guyatt G, Cook DJ; Canadian Critical Care Trials Group. Fluids in Sepsis and Septic Shock (FISSH): protocol for a pilot randomised controlled trial. BMJ Open. 2017 Jul 20;7(7):e017602. doi: 10.1136/bmjopen-2017-017602. PMID 28729329